CLINICAL TRIAL: NCT04583748
Title: Virtual Health Education vs Meditation in Irreversible Age-Related Vision Loss Patients and Their Caregivers: A Pilot Randomized Controlled Trial
Brief Title: Virtual Health Education vs Meditation in Irreversible Age-Related Vision Loss Patients and Their Caregivers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID 19
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: The Art of Living Foundation (Other)
Responsible Party: Principal Investigator, Akshya Vasudev, Consultant Geriatric Psychiatrist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4860
Record Dates: First submitted 2020-09-21; First posted 2020-10-12 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Vision; Disorder, Loss; Caregiver Burnout; Quality of Life; Depression; Anxiety; Sleep
Keywords: Irreversible Age-Related Vision Loss; Caregivers; Quality of Life; Mental Health; Depression; Anxiety; Sleep Quality; Community Integration; Resilience; Caregiver Burden; Sahaj Samadhi Meditation; Health Enhancement Program; Virtual
MeSH Terms: conditions — Caregiver Burden; Depression; Anxiety Disorders; Psychological Well-Being; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Patients will undergo 1:1:1 randomization to Sahaj Samadhi Meditation or Health Enhancement Program or Treatment as Usual, stratified by gender. Twenty-five irreversible age-related vision loss patients and their 25 caregivers will be assigned, on a rolling basis, in the three groups.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will be blinded to the treatment hypothesis, while investigators and treating clinicians will be additionally blinded to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sahaj Samadhi Meditation (Experimental): Participants randomized to the Sahaj Samadhi Meditation (SSM) arm will undergo SSM training in groups of 10. SSM will be delivered virtually using the Cisco WebEx platform by trained, certified non-clinician teachers. Participants will be trained for 4 consecutive days (2 hours/day) in the first week, followed by 1-hour weekly reinforcement sessions for 11 weeks. Participants will also be encouraged to practice twice daily at home for 20 minutes per session. They will be given a daily practice log on which they check off a box indicating if they have done their home practice.
  Interventions: Behavioral: Sahaj Samadhi Meditation
- Health Enhancement Program (Active Comparator): Participants randomized to the Health Enhancement Program (HEP) arm will undergo HEP training in groups of 10. HEP will be delivered virtually using the Cisco WebEx platform by trained non-clinician teachers. Participants will be trained for 4 consecutive days (2 hours/day) in the first week, followed by 1-hour weekly reinforcement sessions for 11 weeks. Participants will also be encouraged to practice twice daily at home for 20 minutes per session. They will be given a daily practice log on which they check off a box indicating if they have done their home practice.
  Interventions: Behavioral: Health Enhancement Program
- Treatment as Usual (No Intervention): Participants randomized to the Treatment as Usual (TAU) arm will continue to receive their treatment as usual. The usual standard of care for irreversible age-related vision patients includes no active treatment since eye surgeons have done all that could possibly be done to restore vision.

INTERVENTIONS:
Behavioral: Sahaj Samadhi Meditation — Sahaj Samadhi Meditation (SSM) is a form of automatic self-transcending meditation that involves relaxed attention to a precise sound (mantra), to allow stress reduction and deep relaxation. This technique is easy to learn and offers the support of a group and facilitator.
  Other Names: SSM
  Arms: Sahaj Samadhi Meditation
Behavioral: Health Enhancement Program — The Health Enhancement Program (HEP) is a standardized program used to teach participants about health promotion, including the benefits of a lifestyle of healthy diet, music, recreation, and exercise. In HEP, participants get the support of a group and facilitator, and talk through and try to implement positive health-enhancing life changes.
  Other Names: HEP
  Arms: Health Enhancement Program

SUMMARY:
Vision loss is common among older adults and leads to an increased risk for depression and difficulties in daily tasks, thus requiring dependence on caregivers. This study will assess the feasibility of providing two virtual interventions, Sahaj Samadhi Meditation (SSM) and Health Enhancement Program (HEP), to supplement care of patients with irreversible age-related vision loss (IARVL) and their caregivers, with the goal of enhancing mental health and quality of life.

DETAILED DESCRIPTION:
Through a high-quality, single-blind, three-arm mixed-method pilot feasibility study using randomized treatment assignment, the study team will assess two new innovative interventions, Sahaj Samadhi Meditation (SSM) and Health Enhancement Program (HEP), both delivered virtually, to augment clinical care of patients with irreversible age-related vision loss (IARVL), with the goal of enhancing mental health and quality of life (QOL) for patients and/or their caregivers. Participants will be blinded to the treatment hypothesis, while investigators and treating clinicians will be additionally blinded to the intervention. Both SSM and HEP will be taught over 4 consecutive days in similar sized groups (10 patients and/or their 10 caregivers) followed by weekly reinforcement sessions for subsequent 11 weeks. Self-rated questionnaires will be used to collect data on quality of life and mental health symptoms at 0-week and 12-week follow-up

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with irreversible age-related vision loss (IARVL) by an experienced ophthalmologist and/or their caregivers.
2. IARVL patients between the age range of 60 to 85 years, while caregivers between the age range of 18 to 85 years.
3. Be able to provide valid informed consent to participate in the research study.
4. Being able to speak as well as understand English without the requirement for interpretation or other communication assistance.
5. Having no significant self-reported or a physician-diagnosed mental health disorder other than depressive and/or anxiety symptoms.
6. Should reach a minimal threshold of depressive and/or anxiety symptoms as confirmed by either a minimum of Centre for Epidemiologic Studies - Depression (CES-D) 20-item scale score of 16 OR a minimum of 8 on the Hospital Anxiety and Depression Scale - Anxiety subscale (HADS-A).
7. Have sufficient hearing to be able to follow verbal instructions
8. Have the ability to sit independently without physical discomfort for 30 minutes.
9. Willing and able to attend virtual intervention via Cisco WebEx software, the four initial training sessions of SSM or HEP and at least 6 out of 11 weekly follow-up sessions.
10. Willing to dedicate 20 minutes twice per day six days per week to their assigned home practice.

Exclusion Criteria:

1. Inability to provide a valid informed consent.
2. Having an underlying major neurocognitive disorder as suggested by a Montreal Cognitive Assessment (MoCA) score < 21.
3. Having significant suicidal ideation as per self-report (CES-D = 3 on item question 14 and/or 15).
4. Having severe depression as confirmed by a CES-D ≥ 24.
5. Participating in other similar studies.
6. Having a lifetime diagnosis of self-reported other serious mental disorders, including bipolar I or II disorder, primary psychotic disorder (schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder).
7. Self-reported substance abuse or dependence within the past 3 months.
8. Having an acutely unstable medical illnesses, including delirium or acute cerebrovascular or cardiovascular events within the last 6 months.
9. Having a terminal medical diagnosis with prognosis of less than 12 months.
10. Having any planned changes to mood-altering medications at the time of enrollment for the next 12 weeks.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-04-09 (Actual); Study Completion 2022-04-09 (Actual)

PRIMARY OUTCOMES:
Number of Potential Participants Approached Per Month | 1 year
  The number of potential participants approached per month will be calculated as a feasibility measure.
Number of Participants who are Successfully Screened | 1 year
  The number of participants who are successfully screened will be calculated as a feasibility measure.
Proportion of Successfully Screened in Participants who Enroll | 1 year
  The proportion of successfully screened in participants who enroll in the study will be calculated as a feasibility measure.
Rate of Retention | 1 year
  The rate of retention of participants in the study will be calculated as a feasibility measure.
Rate of Adherence to Study Protocol | 1 year
  At the end of the study any deviations from the protocol will be examined to determine the rate of adherence to the study protocol. This information will be calculated as a feasibility measure.
Proportion of Planned Ratings that are Completed | 1 year
  The proportion of completed planned ratings will be calculated as a feasibility measure.
Intervention Cost Per Case | 1 year
  The cost per participant of attending the SSM program will be calculated as a feasibility measure.
Percentage of Time Trade-Off (TTO) Questionnaires Completed | 1 year
  The percentage of TTO questionnaires completed by each participant will be examined at the end of the study to assess the completeness of the data as a feasibility measure.
Percentage of Visual Function Index (VF-14) Questionnaires Completed | 1 year
  The percentage of VF-14 questionnaires completed by each participant will be examined at the end of the study to assess the completeness of the data as a feasibility measure.
Percentage of Center for Epidemiologic Studies - Depression (CES-D) Questionnaires Completed | 1 year
  The percentage of CES-D questionnaires completed by each participant will be examined at the end of the study to assess the completeness of the data as a feasibility measure.
Percentage of Hospital Anxiety and Depression Scale - Anxiety (HADS-A) Questionnaires Completed | 1 year
  The percentage of HADS-A questionnaires completed by each participant will be examined at the end of the study to assess the completeness of the data as a feasibility measure.
Percentage of Pittsburgh Sleep Quality Index (PSQI) Questionnaires Completed | 1 year
  The percentage of PSQI questionnaires completed by each participant will be examined at the end of the study to assess the completeness of the data as a feasibility measure.
Percentage of Community Integration Questionnaire (CIQ) Questionnaires Completed | 1 year
  The percentage of CIQ questionnaires completed by each participant will be examined at the end of the study to assess the completeness of the data as a feasibility measure.
Percentage of Connor-Davidson Resilience Scale (CD-RISC) Questionnaires Completed | 1 year
  The percentage of CD-RISC questionnaires completed by each participant will be examined at the end of the study to assess the completeness of the data as a feasibility measure.
Percentage of Zarit Burden Interview (ZBI) Questionnaires Completed | 1 year
  The percentage of ZBI questionnaires completed by each participant will be examined at the end of the study to assess the completeness of the data as a feasibility measure.

SECONDARY OUTCOMES:
Change in Health-Related Quality of Life Score | Weeks 0 and 12
  Change in Health-Related Quality of Life (HRQOL) score as measured by the Time Trade-Off questionnaire (TTO) over a 12-week follow-up. TTO scores range between 0 and 1, with higher scores indicating a higher quality of life.
Change in Vision-Related Quality of Life Score | Weeks 0 and 12
  Change in Vision-Related Quality of Life (VRQOL) score as measured by the Visual Function Index questionnaire (VF-14) over a 12-week follow-up. VF-14 scores range from 0 to 100, with higher scores representing a greater VRQOL.
Change in Depressive Symptoms | Weeks 0 and 12
  Change in depressive symptoms as measured by change in Center for Epidemiologic Studies - Depression (CES-D) scores over a 12-week follow-up. The possible range of CES-D scores is 0 to 60, with the higher scores indicating the presence of more depressive symptomatology.
Change in Anxiety Symptoms | Weeks 0 and 12
  Change in anxiety symptoms as measured by change in Hospital Anxiety and Depression Scale - Anxiety (HADS-A) scores over a 12-week follow-up. Total scores on the HADS-A range from 0 to 21. Higher scores represent higher levels of psychological distress.
Change in Sleep Quality: Pittsburgh Sleep Quality Index (PSQI) | Weeks 0 and 12
  Change in sleep quality as measured by change in Pittsburgh Sleep Quality Index (PSQI) scores over a 12-week follow-up. PSQI scores range from 0 to 21. Higher PSQI scores indicate worse sleep quality.
Change in Community Integration | Weeks 0 and 12
  Change in community integration as measured by change in Community Integration Questionnaire (CIQ) scores over a 12-week follow-up. The overall score for the CIQ ranges from 0 to 29. Higher CIQ score represents greater integration.
Change in Resilience | Weeks 0 and 12
  Change in resilience as measured by change in Connor-Davidson Resilience Scale (CD-RISC) scores over a 12-week follow-up. Total scores for the CD-RISC range from 0 to 40, with higher scores representing greater resilience.
Change in Caregiver Burden | Weeks 0 and 12
  Change in caregiver burden as measured by change in Zarit Burden Interview (ZBI) scores over a 12-week follow-up. Total scores for the ZBI range from 0 to 88. Higher scores represent a more severe self-perceived burden of caregiving.

CONTACTS AND LOCATIONS:
Overall Officials: Akshya Vasudev, MD, Principal Investigator — London Health Sciences Centre; Cindy Hutnik, MD, PhD, Principal Investigator — St. Joseph's Healthcare London

IPD SHARING:
Plan to Share IPD: No